CLINICAL TRIAL: NCT03949361
Title: Glucocorticoid Long-term Administration: Effect on Cold Induced Energy Expenditure and Resting Metabolic Rate
Acronym: GLACIER
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2017-01742
Record Dates: First submitted 2019-04-02; First posted 2019-05-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Thermoregulation Impairment
Keywords: Glucocorticoids; Brown Adipose tissue; Cold Induced Thermogenesis; Resting Metabolic Rate
MeSH Terms: interventions — Skin Temperature; Absorptiometry, Photon; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma Optional biopsy of supraclavicular BAT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients starting glucocorticoids: Patients starting a glucocorticoid therapy measuring primary and secondary endpoints before and after at least 4 weeks of treatment.
  Interventions: Diagnostic Test: Indirect calorimetry; Diagnostic Test: Skin Temperature; Diagnostic Test: Dual energy X-ray Absorptiometry (DXA); Diagnostic Test: Blood Sampling; Diagnostic Test: FDG-PET; Diagnostic Test: Capillary glucose; Diagnostic Test: Biopsy of supraclavicular adipose tissue (optional)
- Patients stopping glucocorticoids: Patients stopping a glucocorticoid therapy measuring primary and secondary endpoints before weaning off glucocorticoids and after a period of at least 3 months.
  Interventions: Diagnostic Test: Indirect calorimetry; Diagnostic Test: Skin Temperature; Diagnostic Test: Dual energy X-ray Absorptiometry (DXA); Diagnostic Test: Blood Sampling; Diagnostic Test: FDG-PET; Diagnostic Test: Capillary glucose; Diagnostic Test: Biopsy of supraclavicular adipose tissue (optional)

INTERVENTIONS:
Diagnostic Test: Indirect calorimetry — Resting energy expenditure
Diagnostic Test: Skin Temperature — Temperature: supraclavicular, infraclavicular, abdominal, mid-thigh, non-dominant lower arm, middle finger tip, left lower leg, left dorsal foot, ear thermometer
Diagnostic Test: Dual energy X-ray Absorptiometry (DXA) — Body composition
Diagnostic Test: Blood Sampling — thyroid-stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), HbA1c, Fibroblast growth factor 21 (FGF21)
Diagnostic Test: FDG-PET — Dynamic PET scanning of the neck-region
Diagnostic Test: Capillary glucose — Prior to fluorodeoxyglucose (FDG)-PET in order to avoid hyperglycemia
Diagnostic Test: Biopsy of supraclavicular adipose tissue (optional) — Ultrasound guided biopsy of the supraclavicular adipose tissue

SUMMARY:
The aim of the study is to investigate whether treatment with glucocorticoids leads to a change in heat production of the human body at mild cold conditions.

DETAILED DESCRIPTION:
Brown adipose tissue (BAT) is a thermogenic tissue that can convert chemical energy directly into heat due to the expression of uncoupling protein 1 (UCP1) protein. Data from preclinical studies shows that glucocorticoids (GCs) inhibit the function of BAT. In clinical practice GCs are often administered due tue their antiinflammatory properties making the investigation of short term (e.g. one week) and long therm (several months) effects practically relevant. This study's objective is to evaluate the effect of glucocorticoid treatment on cold induced thermogenesis (CIT) in humans.

ELIGIBILITY:
Inclusion Criteria:

* Planned therapy with at least 7.5 mg prednisone equivalent per day or higher for more than 28 days (group A)
* Planned weaning off glucocorticoid therapy which lasted al least 28 days with a dosage of at least 7.5 mg prednisone (group B)
* BMI 19-30 kg/m2
* Informed Consent as documented by signature

Exclusion Criteria:

* Insufficient thyroid hormone substitution in case of hypothyroidism
* Uncontrolled diabetes mellitus (HbA1c >7.5%)
* Severe concomitant diseases: chronic heart failure, liver cirrhosis, kidney failure, active cancer
* Known hypersensitivity to cold, e.g. primary or secondary Raynaud's Syndrome
* Known or suspected non-compliance
* Abuse of alcohol or illicit drugs
* Claustrophobia
* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc of the participant
* Previous enrolment into the current study
* Enrolment into another study using ionizing radiation within the previous 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited via the outpatient clinics (endocrinology, rheumathology, ophthalmology, gastroenterology etc.) of the Basel University Hospital.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Cold-induced thermogenesis (CIT) under glucocorticoids | Change from glucocortoid start to +4 to 8 weeks into treatment/ +3 months after weaning off GCs (resp.)
  Comparison of CIT change off-glucocorticoids with warm ischemia time (WIT) on-glucocorticoids by using indirect calorimetry. Comparing two Groups (Observation group A and B) we will address the CIT change from glucocorticoid start to 4-8 weeks into treatment (group A) and the CIT change from glucocorticoid therapy to weaning off upon more than 3 months after glucocorticoid withdrawal (group B)

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | Baseline and +4 to 8 weeks into treatment/ +3 months after weaning off GCs (resp.)
  Comparison of RMR of patients starting GCs or patients stopping GCs, measured by indirect calorimetry
Body composition | Baseline and +4 to 8 weeks into treatment/ +3 months after weaning off GCs (resp.)
  Comparison of body composition concerning muscle mass and fat mass, determined by DXA
Cold stimulated glucose uptake into supraclavicular BAT | Baseline and +4 to 8 weeks into treatment/ +3 months after weaning off GCs (resp.)
  Determination of 'standardized uptake value' (SUV) mean in two volumes of interest on the supraclavicular adipose tissue, after PET-CT
SUV max in supraclavicular adipose tissue depot | Baseline and +4 to 8 weeks into treatment/ +3 months after weaning off GCs (resp.)
  Determination of SUV max in the supraclavicular adipose tissue, after positron emission tomography (PET)-CT

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Matthias, PD Dr. med, Study Director — Klinik Endokrinologie, Diabetes und Metabolismus
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland